CLINICAL TRIAL: NCT03494712
Title: Safety, Tolerability and Pharmacokinetics of S 95010 After Single Escalating Intravenous Doses in Young Healthy Male Subjects. A Randomised, Doubleblind, Placebo-controlled, Monocentre, First-In-Human Study.
Brief Title: Safety of Single Intravenous Administration of S95010 in Human Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CL1-95010-001; 2017-004180-12 (EudraCT Number)
Record Dates: First submitted 2018-02-16; First posted 2018-04-11 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Cardiovascular Diseases
Keywords: healthy volunteer; antimiR; single ascending dose
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- S 95010 (Experimental): Increasing single doses of S 95010 to 5 subjects.
  Interventions: Drug: S 95010
- Placebo (Placebo Comparator): Increasing single doses of Placebo to 2 subjects.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: S 95010 — Single administration of S 95010 in healthy volunteers
  Arms: S 95010
Other: Placebo — Single administration of placebo in healthy volunteers
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess, the safety and tolerability of single ascending doses of S 95010 and to assess the pharmacokinetics (PK) of S 95010.

ELIGIBILITY:
Inclusion Criteria:

* Young healthy male subjects aged between 18 and 45 years (both inclusive)

Exclusion Criteria:

* Any acute or chronic illness or clinically relevant findings such as livers,kidney, spleen, cardiovascular disease, eye disease in the selection/ inclusion visit examinations
* Any abnormal laboratory result on blood and urine samples taken during screening, judged clinically relevant by the investigator
* History of liver dysfunction or total bilirubin or ALT or AST or ALP or γGT > ULN at selection
* History of renal dysfunction or GFR < 75mL/min/1.73 m2 (MDRD equation) at selection

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Safety assessed by incidence of Adverse Events | Through study completion, an average of 12 weeks
  Safety criterion

SECONDARY OUTCOMES:
The PK (pharmacokinetic) profile of S 95010 plasma concentration : Area under the plasma concentration-time curve (AUC) | During Hospitalization Period (Day 1, Day 2, Day 3, Day 4) and during ambulatory follow-up period (at Week 2, Week 4 and Week 12)
  Safety and pharmacokinetic criteria - S 95010 (active parent compound) and its metabolites (if applicable) concentration in serial plasma and urinary samples
The PK profile of S 95010 plasma concentration : Plasma half-life | During Hospitalization Period (Day 1, Day 2, Day 3, Day 4) and during ambulatory follow-up period (at Week 2, Week 4 and Week 12)
  Safety and pharmacokinetic criteria - S 95010 (active parent compound) and its metabolites (if applicable) concentration in serial plasma and urinary samples
The PK profile of S 95010 plasma concentration : Maximum plasma concentration (Cmax) | During Hospitalization Period (Day 1, Day 2, Day 3, Day 4) and during ambulatory follow-up period (at Week 2, Week 4 and Week 12)
  Safety and pharmacokinetic criteria - S 95010 (active parent compound) and its metabolites (if applicable) concentration in serial plasma and urinary samples

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Clinical Pharmacology Unit - Stuivenberg Hospital, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Researchers can ask for a study protocol, patient-level and/or study-level clinical trial data including clinical study reports (CSRs).
  They can ask all interventional clinical studies:
  * submitted for new medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier or an affiliate are the Marketing Authorization Holders (MAH). The date of the first Marketing Authorization of the new medicine (or the new indication) in one of the EEA Member States will be considered within this scope.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: study-level clinical trial data — https://clinicaltrials.servier.com/